CLINICAL TRIAL: NCT02581280
Title: Population Pharmacokinetics of Teicoplanin, Levofloxacin, Piperacillin/Tazobactam, Meropenem, Vancomycin, Remifentanil, Cefepime, Cefpirome, Sufentanil, Midazolam, Clopidogrel, Ticagrelor, Prasugrel During Veno-arterial Extracorporeal Membrane Oxygenation (VA ECMO)
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0919
Record Dates: First submitted 2015-10-08; First posted 2015-10-20 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Cardiac Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Residual blood samples(1~2 cc) at each sampling time are collected from all subjects while using ECMO for drug concentration assays(LC-MS/MS etc.). After ECMO device is removed, residual arterial blood samples(1~2 mls) at each sampling time are collected and drug concentrations are assayed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- On ECMO: patients who are concomitantly receiving teicoplanin or levofloxacin or piperacillin/tazobactam or meropenem or vancomycin or remifentanil or cefepime or cefpirome or sufentanil or midazolam or clopidogrel or ticagrelor or prasugrel during ECMO
  Interventions: Other: Residual blood
- Off ECMO: patients who are concomitantly receiving teicoplanin or levofloxacin or piperacillin/tazobactam or meropenem or vancomycin or remifentanil or cefepime or cefpirome or sufentanil or midazolam or clopidogrel or ticagrelor or prasugrel after removing ECMO
  Interventions: Other: Residual blood

INTERVENTIONS:
Other: Residual blood — Residual blood samples(1~2 cc) at each sampling time are collected from all subjects while using ECMO for drug concentration assays(LC-MS/MS etc.).

SUMMARY:
Extracorporeal membrane oxygenation (ECMO) is the device which increases the supply of oxygen to the body tissues in vitro and to assist in heart and lung function. Venoarterial (VA) ECMO is used in patients with cardiogenic shock, cardiac arrest, ventricular arrhythmia and is able to secure a time to self-recovery by reducing the excessive stimulation applied to the heart. However, in ECMO patients, pharmacokinetics of drugs are changing such as increased volume of distribution (Vd) or decreased clearance (CL). For this reason, it is hard to provide the best treatment in ECMO patients. The study is to evaluate whether the PK of drugs is influenced by VA ECMO and to recommend the optimal dosing strategies for proposed drugs in adult patients receiving VA ECMO.

ELIGIBILITY:
Inclusion Criteria:

* patient who are ≥ 19 years old and receiving VA ECMO in Severance Hospital, Yonsei University Health System.
* patient who are receiving one of these drugs: teicoplanin or levofloxacin or piperacillin/tazobactam or meropenem or vancomycin or remifentanil or cefepime or cefpirome or sufentanil or midazolam or clopidogrel or ticagrelor or prasugrel
* patients who are agreed to participate in this study

Exclusion Criteria:

* patients who are pregnant
* patients who are receiving drugs that could affect study drug's concentration due to drug-drug interaction.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 19 who are receiving teicoplanin or levofloxacin or piperacillin/tazobactam or remifentanil or sufentanil or clopidogrel or ticagrelor while using VA ECMO in Severance Hospital, Yonsei University Health System.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2014-12; Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Serum or plasma concentration | Between day0 to day3 after removing ECMO
  Serum or plasma concentration of teicoplanin or levofloxacin or piperacillin/tazobactam or meropenem or vancomycin or remifentanil or cefepime or cefpirome or sufentanil or midazolam or clopidogrel or ticagrelor or prasugrel
Pharmacokinetic parameter: Cmax | Between day0 to day3 after removing ECMO
Pharmacokinetic parameter: Tmax | Between day0 to day3 after removing ECMO
Clearance | Between day0 to day3 after removing ECMO
volume of distribution | Between day0 to day3 after removing ECMO
absorption rate constant | Between day0 to day3 after removing ECMO
  absorption rate constant (if the drug is orally administered),
elimination half life | Between day0 to day3 after removing ECMO
area under the curve (AUC) | Between day0 to day3 after removing ECMO
  area under the curve (AUC) (if possible)

CONTACTS AND LOCATIONS:
Overall Officials: Jin Wi, MD, Principal Investigator — Severance Hospital
Locations (1):
- Division of Cardiology, Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Kim H, Jin BH, Yang S, Hahn J, Kang S, Kim D, Lee H, Kwack H, Chae SU, Bae SK, Wi J, Chang MJ. Effect of Extracorporeal Membrane Oxygenation Flow Rate on Midazolam Clearance: A Population Pharmacokinetic Study. Anesthesiology. 2026 Feb 1;144(2):485-488. doi: 10.1097/ALN.0000000000005811. Epub 2025 Nov 25. No abstract available. PMID 41325279
- [Derived] Hahn J, Min KL, Kang S, Yang S, Park MS, Wi J, Chang MJ. Population Pharmacokinetics and Dosing Optimization of Piperacillin-Tazobactam in Critically Ill Patients on Extracorporeal Membrane Oxygenation and the Influence of Concomitant Renal Replacement Therapy. Microbiol Spectr. 2021 Dec 22;9(3):e0063321. doi: 10.1128/Spectrum.00633-21. Epub 2021 Dec 22. PMID 34937189
- [Derived] Kang S, Jang JY, Hahn J, Kim D, Lee JY, Min KL, Yang S, Wi J, Chang MJ. Dose Optimization of Cefpirome Based on Population Pharmacokinetics and Target Attainment during Extracorporeal Membrane Oxygenation. Antimicrob Agents Chemother. 2020 Apr 21;64(5):e00249-20. doi: 10.1128/AAC.00249-20. Print 2020 Apr 21. PMID 32122899
- [Derived] Hahn J, Yang S, Min KL, Kim D, Jin BH, Park C, Park MS, Wi J, Chang MJ. Population pharmacokinetics of intravenous sufentanil in critically ill patients supported with extracorporeal membrane oxygenation therapy. Crit Care. 2019 Jul 9;23(1):248. doi: 10.1186/s13054-019-2508-4. PMID 31288863
- [Derived] Wi J, Noh H, Min KL, Yang S, Jin BH, Hahn J, Bae SK, Kim J, Park MS, Choi D, Chang MJ. Population Pharmacokinetics and Dose Optimization of Teicoplanin during Venoarterial Extracorporeal Membrane Oxygenation. Antimicrob Agents Chemother. 2017 Aug 24;61(9):e01015-17. doi: 10.1128/AAC.01015-17. Print 2017 Sep. PMID 28674057